CLINICAL TRIAL: NCT04641364
Title: Safety and Tolerance Study of Recombinant Human Albumin Injection in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ART-2019-001
Record Dates: First submitted 2020-10-12; First posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-09

CONDITIONS: Ascites
MeSH Terms: conditions — Ascites | interventions — Sodium Chloride; Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control: placebo (Placebo Comparator): Subjects received 0.9% sodium chloride injection.
  Interventions: Drug: Placebo
- Control: Human Serum Albumin(HSA) (Active Comparator): Subjects received Human Serum Albumin, 10 g for each day, three days for a cycle, and totally three cycles.
  Interventions: Drug: human albumin injection
- Experimental:recombinant human albumin (Experimental): Subjects received recombinant Human Serum Albumin, 1.25g, 5g, 10g, 20g, 30 g for the single dose study. For the multiple dose study, subjects received recombinant Human Serum Albumin, 10 g for each day, three days for a cycle, and totally three cycles.
  Interventions: Drug: recombinant human albumin injection

INTERVENTIONS:
Drug: recombinant human albumin injection — single dose or multiple doses of intravenous infusion
  Other Names: Intravenous infusion of recombinant human albumin injection
  Arms: Experimental:recombinant human albumin
Drug: Placebo — Single dose intravenous infusion of 0.9% sodium chloride injection
  Other Names: Intravenous infusion of 0.9% sodium chloride injection
  Arms: Control: placebo
Drug: human albumin injection — multiple doses of intravenous infusion
  Other Names: Intravenous infusion of human albumin injection
  Arms: Control: Human Serum Albumin(HSA)

SUMMARY:
A phase I, single-center, randomized, double-blind, placebo-controlled single dose escalation study, and a positive-controlled multiple dose extension study to evaluate the safety, tolerance, pharmacokinetics and immunogenicity of recombinant human albumin injection in healthy subjects

DETAILED DESCRIPTION:
This study was to evaluate the safety, tolerability, pharmacokinetics and immunogenicity of recombinant human albumin injection in healthy volunteers. The safety, tolerance, pharmacokinetics and immunogenicity of recombinant human albumin injection were evaluated in a single center, randomized, double-blind, placebo-controlled single dose incremental trial in healthy volunteers. The study was divided into two stages: the first stage was a single dose and dose increasing stage (including 5 dose groups with increasing dose, and each group was set with placebo control); the second stage was multiple administration stage (with positive control). The safety, tolerance, pharmacokinetics, immunogenicity and other early clinical data of recombinant human albumin were collected and analyzed in the two stages. The initial dose was 1.25g. The highest dose group was set at 30g. The dose groups of 1.25, 5, 10, 20 and 30 g / time were preset in the single dose stage (dose increasing stage). The dosage was 10 g / Day in multiple administration stage.

ELIGIBILITY:
Inclusion Criteria:

1）Informed consent form signed; 2) To be able to complete the study; 3) Subjects (including partners) are willing to take contraceptive measures; 4) 18-55 years of age; 5) Male subjects are no less than 50 kg.Female subjects are no less than 45 kg. Body mass index is 18-28kg / m2; 6) Normal cardiac function, defined as left ventricular ejection fraction (LVEF) ≥ 50%; 7) Physical examination and vital signs are normal.

Exclusion Criteria:

1. Cigarettes Smoking subjects.
2. Allergic constitution (multiple drugs and food allergies);
3. History of drug use and/or alcohol abuse;
4. Blood donation or massive blood loss (> 450 mL) within three months before screening;
5. Taking any drugs, prescription, over-the-counter, vitamin products or herbal medicine within 14 days before screening;
6. Diet or exercise have changed recently;
7. Using study drugs within three months;
8. Risk of bleeding, such as hemorrhoids, acute gastritis or stomach and duodenal ulcers;
9. ECG abnormalities (QTc > 470ms for males, > 480ms for females);
10. Female subjects are in lactation. Pregnancy test is positive;
11. Other Clinical laboratory tests abnormalities;
12. Viral screening test is positive, including HBV, HCV, HIV, and Treponema pallidum;
13. Developing Acute disease;
14. Eating chocolate, any caffeine-containing or jaundice-rich food or drink 24 hours prior to the use of the study drug;
15. Taking any alcoholic products. Alcohol test is positive..
16. Drug test is positive. History of drug abuse or drug use in the past five years;
17. Inability for intravenous injection or blood collection;
18. Using biological products (including live vaccines) within the last 3 months. Planing to use vaccines during the study period. Having received corticosteroid or human plasma product system treatment within 1 month.
19. Renal function is abnormal, glomerular filtration rate <80 mL/min (according to the simplified MDRD formula);
20. History of glaucoma, eye disease.
21. History of cancer or other serious systemic diseases, especially heart, liver, kidney, digestive tract, nervous system, metabolic abnormalities, immune abnormalities or mental disorders;
22. History of immunodeficiency or hypofunction;
23. Received major surgery within 2 years.
24. Other subjects by investigator opinion..

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerance | Day 1-Day 57 for single doses study. Day 1-Day 106 for multiple doses study.
  AE

SECONDARY OUTCOMES:
PK parameters | Day 1-Day 57 for single doses study. Day 1-Day 106 for multiple doses study.
  Maximum Plasma Concentration（Cmax）
PK parameters | Day 1-Day 57 for single doses study. Day 1-Day 106 for multiple doses study.
  time to Maximum Plasma Concentration（Tmax）
PK parameters | Day 1-Day 57 for single doses study. Day 1-Day 106 for multiple doses study.
  half life (t1/2）
Pharmacodynamic parameters | Day 1-Day 57 for single doses study. Day 1-Day 106 for multiple doses study.
  Red blood cell specific volume
Pharmacodynamic parameters | Day 1-Day 57 for single doses study. Day 1-Day 106 for multiple doses study.
  Plasma colloid osmotic pressure
Immunogenicity | Day 1-Day 57 for single doses study. Day 1-Day 106 for multiple doses study.
  Percentage of patients with positive reaction

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, Dr, Study Director — The first affiliated hospital of Jilin University
Locations (1):
- the first hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No